CLINICAL TRIAL: NCT01515735
Title: Evaluation of LOXL1 Polymorphism in Pseudoexfoliation Syndrome in the Korean Population
Brief Title: LOXL1 Polymorphism in Pseudoexfoliation Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2011-06-035
Record Dates: First submitted 2012-01-18; First posted 2012-01-24 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Pseudoexfoliation Syndrome
MeSH Terms: conditions — Exfoliation Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pseudoexfoliation: The study group composted of the patients with pseudoexfoliation syndrome

SUMMARY:
To evaluate the association profiles of the lysyl oxidase-like 1 gene polymorphisms with pseudoexfoliation syndrome in the Korean population, Genotypes of lysyl oxidase-like 1 gene were analyzed by direct sequencing.

DETAILED DESCRIPTION:
To evaluate the association profiles of the lysyl oxidase-like 1 gene polymorphisms with pseudoexfoliation syndrome in the Korean population, peripheral blood sampling will be done from the patients with pseudoexfoliation.

And genotypes of the three single nucleotide polymorphisms of lysyl oxidase-like 1 gene , rs1048661, rs3825942, rs2165241 were analyzed by direct sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Pseudoexfoliation

Exclusion Criteria:

* medical condition that peripheral blood sampling cannot be done

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the groups or cohorts will be recruited from glaucoma clinic in Samsung medical center
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Genotypes of the three single nucleotide polymorphisms of LOXL1 (rs1048661, rs3825942, rs2165241) | about 1 year (when all patients were recruited)
  Genotypes of the three single nucleotide polymorphisms of LOXL1 were analyzed by direct sequencing, after obtained from the peripheral blood sampling from patients.

CONTACTS AND LOCATIONS:
Overall Officials: Changwon Kee, M.D., PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, South Korea

REFERENCES:
- [Result] Mori K, Imai K, Matsuda A, Ikeda Y, Naruse S, Hitora-Takeshita H, Nakano M, Taniguchi T, Omi N, Tashiro K, Kinoshita S. LOXL1 genetic polymorphisms are associated with exfoliation glaucoma in the Japanese population. Mol Vis. 2008 Jun 5;14:1037-40. PMID 18552979
- [Result] Fuse N, Miyazawa A, Nakazawa T, Mengkegale M, Otomo T, Nishida K. Evaluation of LOXL1 polymorphisms in eyes with exfoliation glaucoma in Japanese. Mol Vis. 2008 Jul 21;14:1338-43. PMID 18648524